CLINICAL TRIAL: NCT04057521
Title: Coordinated HEalthcare for Complex Kids Impact on Medicaid Expenditures
Brief Title: Coordinated HEalthcare for Complex Kids
Acronym: CHECK
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Centers for Medicare and Medicaid Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Benjamin Van Voorhees, MD, MPH, Professor of Pediatrics, University of Illinois at Chicago
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2014-0738
Record Dates: First submitted 2019-08-09; First posted 2019-08-15 (Actual); Last update posted 2019-08-15 (Actual); Status verified 2019-08

CONDITIONS: Asthma; Diabetes Mellitus; Sickle Cell Disease; Premature Birth
Keywords: care coordination; Children; Young adults; Chronic disease
MeSH Terms: conditions — Asthma; Diabetes Mellitus; Anemia, Sickle Cell; Premature Birth; Chronic Disease

STUDY DESIGN:
Intervention Model Description: For the purpose of program evaluation; 6,259 participants who met eligibility criteria for CHECK were randomized. These participants had no previous exposure to CHECK and were randomized to either enrollment into the CHECK program or to usual care (comparison group). Purposive randomization to CHECK or usual care by age, disease and risk level was conducted by Mathmatica.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CHECK Program (Experimental): Participants were offered enrollment into CHECK care coordination services.
  Interventions: Other: Care Coordination
- Comparison Group (Active Comparator): Participants were not offered enrollment into CHECK.
  Interventions: Other: Care Coordination

INTERVENTIONS:
Other: Care Coordination — Comprehensive care coordination.
  Other Names: Demonstration project

SUMMARY:
The University of Illinois Health and Health Sciences System (UI Health) developed an integrated care management quality improvement model designed to provide comprehensive care coordination for Medicaid insured minority children and young adults with chronic health conditions living in Chicago. This program, called CHECK (Coordinated HEalthcare for Complex Kids), targeted children and young adults with chronic disease.

DETAILED DESCRIPTION:
The University of Illinois Health and Health Sciences System (UI Health) developed an integrated care management quality improvement model designed to provide comprehensive care coordination for Medicaid insured minority children and young adults with chronic health conditions living in Chicago. This program, called CHECK (Coordinated HEalthcare for Complex Kids), was funded by a Centers for Medicare and Medicaid Services Innovation (CMMI) Award. The CHECK model took a broad approach to health promotion by addressing social determinants of health, caregiver wellness and mental health needs; in addition to disease management. The program targeted children and young adults from birth to age 25 with diagnoses of asthma, diabetes, sickle cell disease, seizure disorder or prematurity. All participants were enrolled in either the traditional (fee-for-service) state Medicaid program or a Medicaid Managed Care Organization (MCO) in Illinois. CHECK provided access to care coordination delivered by community health workers; mental health services and health education.

CHECK was designed as a demonstration program and participants were enrolled passively over time and received different services depending on their level of risk and need. One primary aim of the CHECK program was to decrease Medicaid expenditures over a three-year period by decreasing unnecessary emergency department visits and hospitalizations.

Though CHECK was designed as a care delivery demonstration program, in April, 2016 we had the opportunity to prospectively randomize 6,259 participants who met eligibility criteria for CHECK, for the purpose of program evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Age 0-25 years;
* Documentation of asthma,
* Diabetes mellitus (type 1 or 2), sickle cell disease,
* Seizure disorder or
* Prematurity; 3)
* Enrolled in Medicaid; and
* Ride in Cook County, Illinois.

Exclusion criteria:

• None

Max Age: 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6259 (Actual)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-08-31 (Actual); Study Completion 2018-08-31 (Actual)

PRIMARY OUTCOMES:
Annual inpatient healthcare utilization per 1000 patient years | Three years
  Number of inpatient hospitalizations/1000 patient years obtained from the Illinois Medicaid paid claims for CHECK participants using the Care Coordination Claims Data (CCCD) provided by the Illinois Department of Healthcare and Family Services (HFS).Claims for the same patient identifier with overlapping service dates were considered one hospitalization. Due to the fact that professional service claims may be submitted independent from facility claims, those claims with the same patient identification number, national provider ID (NPI), and service date were considered the same event to avoid duplication.
Annual emergency room healthcare utilization per 1000 patient years | Three years
  Number of emergency room visits/1000 patient years obtained from the Illinois Medicaid paid claims for CHECK participants using the Care Coordination Claims Data (CCCD) provided by the Illinois Department of Healthcare and Family Services (HFS). The number of inpatient hospitalizations per patient were identified using inpatient facility claims. The number of ED visits per patient were identified from outpatient facility claims or professional claims with revenue codes indicating an ED place of service or Current Procedural Terminology (CPT) codes for emergency services. Due to the fact that professional service claims may be submitted independent from facility claims, those claims with the same patient identification number, national provider ID (NPI), and service date were considered the same event to avoid duplication.
Annual outpatient visit healthcare utilization per patient per 1000 patient years | Three years
  Number of outpatient visits/1000 patient years obtained from the Illinois Medicaid paid claims for CHECK participants using the Care Coordination Claims Data (CCCD) provided by the Illinois Department of Healthcare and Family Services (HFS).Outpatient visits were defined as outpatient facility claims or professional service claims with evaluation and management CPT codes for office visits (excluding observation or outpatient surgery).Due to the fact that professional service claims may be submitted independent from facility claims, those claims with the same patient identification number, national provider ID (NPI), and service date were considered the same event to avoid duplication.

SECONDARY OUTCOMES:
Annual inpatient healthcare expenditures per patient | Three years
  Annual inpatient healthcare expenditures are reported as expenditures/patient/year (US dollars).For the inpatient visit expenditures, costs associated with any remaining outpatient or professional claims with overlapping dates of service were considered part of the event.
Annual emergency room healthcare expenditures per patient | Three years
  Annual emergency room healthcare expenditures are reported as expenditures/patient/year (US dollars).For the emergency room visit expenditures, costs associated with any remaining outpatient or professional claims with overlapping dates of service were considered part of the event.
Annual outpatient healthcare expenditures per patient | Three years
  Annual outpatient healthcare expenditures are reported as expenditures/patient/year (US dollars). Outpatient visits were defined as outpatient facility claims or professional service claims with evaluation and management CPT codes for office visits (excluding observation or outpatient surgery).
Annual prescription healthcare expenditures per patient | Three years
  Annual prescription healthcare expenditures are reported as expenditures/patient/year (US dollars). Prescription expenditures were obtained from the prescription drug file of the CCCD.
Annual "other" healthcare expenditures per patient | Three years
  Annual "other" healthcare expenditures are reported as expenditures/patient/year (US dollars). Expenditures not attributable to inpatient, ED, outpatient visits, or prescription costs were considered 'other' and include services such as observation, outpatient surgery, dental, mental health, labs, and radiology.
Annual total healthcare expenditures per patient | Three years
  Annual total healthcare expenditures are reported as expenditures/patient/year (US dollars). Expenditures were measured for each patient overall, and by category of service (e.g., inpatient, ED, outpatient visits, prescriptions, and other). Outpatient visits were defined as outpatient facility claims or professional service claims with evaluation and management CPT codes for office visits (excluding observation or outpatient surgery). Prescription expenditures were obtained from the prescription drug file of the CCCD. For the inpatient, ED, and outpatient visit expenditures, costs associated with any remaining outpatient or professional claims with overlapping dates of service were considered part of the event. Total expenditures per patient were defined as the sum of all paid claims for any covered service - (e.g., inpatient, ED, outpatient visits, prescriptions, and other).

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin VanVoorhees, MD, Principal Investigator — University of Illinois at Chicago

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Glassgow AE, Martin MA, Caskey R, Bansa M, Gerges M, Johnson M, Marko M, Perry-Bell K, Risser HJ, Smith PJ, Van Voorhees B. An innovative health-care delivery model for children with medical complexity. J Child Health Care. 2017 Sep;21(3):263-272. doi: 10.1177/1367493517712063. Epub 2017 Jun 5. PMID 29119824
- [Background] Bansa M, Glassgow AE, Martin M, Caskey R, Paulson A, Minier M, Roper P, Mitacek R, Wilder J, Van Voorhees B. Development of a Community-Based Medical Neighborhood for Children with Chronic Conditions. Prog Community Health Partnersh. 2019;13(1):83-95. doi: 10.1353/cpr.2019.0011. PMID 30956250
- [Derived] Caskey R, Moran K, Touchette D, Martin M, Munoz G, Kanabar P, Van Voorhees B. Effect of Comprehensive Care Coordination on Medicaid Expenditures Compared With Usual Care Among Children and Youth With Chronic Disease: A Randomized Clinical Trial. JAMA Netw Open. 2019 Oct 2;2(10):e1912604. doi: 10.1001/jamanetworkopen.2019.12604. PMID 31584682